CLINICAL TRIAL: NCT06007027
Title: Vaginal Laser Therapy for Genitourinary Syndrome in Breast Cancer Survivors - A Randomized, Blinded, Placebo-controlled Study
Brief Title: Vaginal CO2 Laser Therapy for Genitourinary Syndrome in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VagLaser
Record Dates: First submitted 2023-08-01; First posted 2023-08-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: laser; mamma cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active laser group (Experimental): In the active laser group, participants are treated intravaginally with the fractional microablative CO2 laser system (SmartXIDE2V2LR, MonaLisa Touch, DEKA, Florence, Italy), using the following setting; dot power 30 watt, dwell time 1000 μs, dot spacing 1000 μs and the smart stack parameter from 2 to 3. At the level of the vaginal introitus, the dot power decreases to 20 Watt.
  Interventions: Device: SmartXIDE2V2LR, Monalisa Touch, DEKA, Florence, Italy
- Sham laser group (Sham Comparator): In the sham laser group, participants are treated intravaginally with the fractional microablative CO2 laser system (SmartXIDE2V2LR, Monalisa Touch, DEKA, Florence, Italy), using the following setting; dot power 0,5 watt, dwell time 100 μs, dot spacing 2000 μs and the smart stack parameter from 1 to 1
  Interventions: Device: SmartXIDE2V2LR, Monalisa Touch, DEKA, Florence, Italy

INTERVENTIONS:
Device: SmartXIDE2V2LR, Monalisa Touch, DEKA, Florence, Italy — The laser probe is gently inserted up to the top of the vagina, and subsequently withdrawn and rotated in order to deliver a complete treatment of the vaginal wall.

SUMMARY:
This project will be based on three studies over a period on three years. The first study is a dose response study that includes 30 breast cancer survivors. They will receive a total of 5 laser treatments with 4-6 weeks intervals The second study is a double-blind randomized controlled trial, that includes 60 breast cancer survivors. 30 of those will receive active intervention and 30 will receive placebo laser treatment and act as controls. Based on the results of the dose response study, a treatment consists of three to five laser treatments every 3 weeks. The third and last study is a one-year follow-up on study two. The conditions are evaluated before and after each treatment by questionnaires, vaginal fluid pH values, punch biopsies and vaginal and urine microbiome. The studies is conducted at the Department of Obstetrics and Gynaecology at Randers Regional Hospital in collaboration with Department of Obstetrics and Gynaecology and Department of Oncology at Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivor in endocrine therapy
* Symptomatic genitourinary symdrom of menopause with vaginal discomfort and/or dyspareunia
* Able to read and understand Danish
* Able to give written informed consent

Exclusion Criteria:

* Pelvic organ prolapse ≥ stage 2 according to the Pelvic Organ Prolapse Quantification staging system
* Use of non-hormonal/hormonal vaginal therapies (1 and 12 months prior to the baseline visit, respectively)
* Use of Chemotherapy (6 months prior to the baseline visit)
* Acute urinary tract infection or active genital infection
* History of vaginal reconstructive surgery

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Vaginal dryness | Symptom data is collected at baseline visit and one month after the last treatment
  Participant are asked to complete the 10-cm visual analog scale (VAS) ranging for 0 to 10, with higher score indicating worse vaginal dryness.

SECONDARY OUTCOMES:
Change in vaginal pain, itching and soreness | Symptom data is collected at baseline visit and one month after the last treatment
  Evaluated with visual analog scale for vaginal pain, itching, soreness. 10-cm visual analog scale (VAS) ranging for 0 to 10, with higher score indicating worse symptoms.
Female Sexual Function Index | Symptom data is collected at baseline visit and one month after the last treatment
  Sexual function parameters; desire, arousal, lubrication, orgasm, satisfaction and pain. Range 2-36, the threshold of 26.55 indicates sexual dysfunction
Sexual complaint screener - women | Symptom data is collected at baseline visit and one month after the last treatment
  Addressing all domains of sexual dysfunction. Range 0-60, higher score indicate increased symptom severity
Urogenital Distress Inventory | Symptom data is collected at baseline visit and one month after the last treatment
  For urinary symptoms; irritative symptoms, obstructive/discomfort and stress symptoms. Range 0-18, higher score indicate higher disability
International Consultation on Incontinence Questionnaire Female Urinary Tract Symptoms Sex | Symptom data is collected at baseline visit and one month after the last treatment
  Evaluation of female sexual matters associated with their lower urinary tract symptoms. Range 0-14, higher values indicating increased symptom severity.
Vaginal health index | Vaginal health index is evaluated at baseline visit and one month after the last treatment
  subjective scoring of moisture, fluid volume, epithelial integrity and elasticity and objective scoring of pH. Range 5-25, higher scores indicate better health
Vaginal biopsy | Vaginal biopsy is collected at baseline visit and one month after the last treatment
  The biopsy of 4*4 mm is taken from the lateralt vaginal wall, 2-3 cm from inotroitus. Afterwards fixated i formalin and the processed for light microsopy by a specialized gynaecological pathologist reporting on the changes in the histology of vaginal epithel and lamina propria.
Vaginal and urinary microbiota | Vaginal and urine microbiota are collected at baseline visit and one month after the last treatment
  One polyester swap (FLOQSwab) is used to sample mid-vagina for microbial analysis and immediately been placed at - 80 °C until further processing. Urine is collected in a 50 mL collection tube using the clean catch method for women. Afterwards aliquoted into 10 mL fractions and immediately been placed at - 80 °C until further processing.
  DNA is isolated from samples using standard DNA isolation kits and microbiota composition determined using 16S rRNA gene sequencing. Microbiota composition is compared between groups and over time based on alpha- and beta-diversity measures, as well as changes in relative abundances of individual bacteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jacobsen S, Bennetsen MH, Nielsen PS, Glavind-Kristensen M, Jensen AB, Forman A, Waldstrom M, Bor P. Impact of fractional CO2 laser therapy on vaginal wall histology in breast cancer survivors. Lasers Med Sci. 2026 Feb 10;41(1):26. doi: 10.1007/s10103-026-04829-0. PMID 41665827
- [Derived] Jacobsen S, Glavind-Kristensen M, Jensen AB, Forman A, Bor P. Vaginal CO2 laser therapy for genitourinary syndrome in breast cancer survivors-VagLaser study protocol: a randomized blinded, placebo-controlled trial. BMC Cancer. 2023 Nov 29;23(1):1164. doi: 10.1186/s12885-023-11656-x. PMID 38031020